CLINICAL TRIAL: NCT06903026
Title: PRevalence Of Transient Global Amnesia in Obstructive Sleep Apnea Syndrome
Acronym: PROTOS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8781
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Transient Global Amnesia
Keywords: Transient Global Amnesia; Sleep apnea syndrome
MeSH Terms: conditions — Amnesia, Transient Global; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Amnesic stroke is an amnestic syndrome lasting less than 24 hours characterized by the occurrence of anterograde amnesia often associated with retrograde amnesia, the pathophysiology of which is still poorly understood at present. A recent study on a small sample size (N=29) highlighted an association between obstructive sleep apnea syndrome and amnesic stroke. Our study seeks to confirm or refute these results on a larger cohort (N=200-250). A better understanding of the pathophysiological processes involved would open up new therapeutic avenues.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients seen for consultation in the Neuropsychology Department of Strasbourg University Hospital between March 1, 2015 and December 31, 2021 following an episode of amnestic stroke meeting the Hodges and Warlow criteria:
* The stroke must have been documented and reported by a competent witness present during the stroke.
* Anterograde amnesia during the stroke.
* Absence of vigilance, personality, and cognitive disorders other than memory disorders (aphasia, apraxia, etc.).
* Absence of focal neurological symptoms during the episode and its aftermath.
* Absence of epileptic manifestations.
* Resolution of the episode in less than 24 hours.
* Exclusion of patients with a history of recent head trauma or active epilepsy (undergoing regular treatment or having experienced a seizure in the last 2 years).
* Subjects who have not expressed opposition to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Patients who have expressed opposition to the retrospective reuse of their data for scientific research purposes.
* Patients with active epilepsy
* Patients with recent head trauma
* Patients with an MMS < or equal to 25
* Subject under guardianship or curatorship
* Subject under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients seen for consultation in the Neuropsychology Department of Strasbourg University Hospital between March 1, 2015 and December 31, 2021 following an episode of amnestic stroke meeting the Hodges and Warlow criteria.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of obstructive sleep apnea syndrome in patients who have experienced an amnestic stroke. | Within the last 2 years
  Presence or absence of obstructive sleep apnea syndrome reported by a witness present during the stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neurologie - CHU de Strasbourg - France, Strasbourg, France